CLINICAL TRIAL: NCT05844020
Title: Assessment of Survivor and Provider Perceptions of Trauma and Violence Informed Care Among Black Women
Brief Title: Perceptions of Trauma and Violence Informed Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: Matthew Walker Comprehensive Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-05-1198
Record Dates: First submitted 2023-03-14; First posted 2023-05-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Intimate Partner Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TVIC Intervention (Experimental)
  Interventions: Behavioral: Educational materials
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Educational materials — Trauma-informed intimate partner violence screening, brief interventions, and referrals to treatment by providers
  Arms: TVIC Intervention

SUMMARY:
The purpose of this study is to adapt, implement and evaluate a trauma and violence informed care intervention designed for Black women in middle Tennessee.

DETAILED DESCRIPTION:
The primary goal is the adaptation, implementation and evaluation of a trauma and violence informed care (TVIC) intervention designed for Black women in middle Tennessee. In this 5-year RCMI project, the investigators propose 3 aims. Aim 1) Engage a stakeholder committee of patients, providers, and experts (COPE) to adapt a TVIC intervention for Black women and their healthcare providers at Meharry. [Years 1-2]. Aim 2) Implement and prospectively evaluate the adapted TVIC intervention at the healthcare provider-level, measuring changes in Meharry healthcare provider's self-efficacy for TVIC implementation and alignment with TIC knowledge, attitudes, and practices. [Years 2-3] Aim 3) Implement the adapted TVIC intervention at the patient-level to provide trauma-informed IPV screening, brief interventions, and referrals to treatment (SBIRT), and rigorously evaluate this TVIC intervention's impact on the primary outcome of patient-perceived usefulness of intervention and reported linkage to IPV services, and the secondary outcome of changes at the clinic-level relative to climate and culture, through a non-randomized pragmatic trial design. [Year 4-5].

ELIGIBILITY:
Inclusion Criteria:

* Meharry or Matthew Walker Comprehensive Health Center female patients
* Self-identify as Black
* Self-identify as intimate partner violence survivors
* English or Spanish language fluency

Exclusion Criteria:

* Not Black female intimate partner violence survivor of Meharry or Matthew Walker Comprehensive Health Center
* Those without English or Spanish language fluency

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who received appropriate intimate partner violence screening and trauma/mental health services referral | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No